CLINICAL TRIAL: NCT00829309
Title: A Relative Bioavailability Study of 80 mg Pravastatin Sodium Tablets Under Non-Fasting Conditions
Brief Title: Pravastatin 80 mg Tablets Dosed in Healthy Subjects Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R05-0202
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pravastatin (Experimental): Pravastatin 80 mg Tablet (test) dosed in first period followed by Pravachol® 80 mg Tablet (reference) dosed in second period
  Interventions: Drug: Pravastatin
- Pravachol® (Active Comparator): Pravachol® 80 mg Tablet (reference) dosed in first period followed by Pravastatin 80 mg Tablet (test) dosed in second period
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — 80 mg Tablet
  Arms: Pravastatin
Drug: Pravastatin — 80 mg Tablets
  Other Names: Pravachol® 80 mg Tablets
  Arms: Pravachol®

SUMMARY:
This study compared the relative bioavailability (rate and extent of absorption) of Pravastatin Sodium Tablets 80 mg by Teva Pharmaceutical Industries, Ltd. with that of Pravachol® Tablets 80 mg by Bristol-Myers Squibb Company following a single oral dose (1 x 80 mg tablet)in healthy adult male subjects administered under non-fasting conditions.

DETAILED DESCRIPTION:
Detailed Description

Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

Outcome: Confidence interval fell within 80-125% therefore met the FDA Bioequivalence criteria; no drug related, serious, unexpected adverse events were reported during the study.

ELIGIBILITY:
Inclusion Criteria

* Screening Demographics: All subjects selected for this study will be healthy men 18 years of age or older at the time of dosing.
* The subject's body mass index (BMI) should be less than or equal to 30.
* Screening Procedures: Each subject will complete the screening process within 28 days prior to period I dosing.
* Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed and signed by each potential participant before full implementation of screening procedures.
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature.
* The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.
* The screening clinical laboratory procedures will include:

  * HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count
  * CLINICAL CHEMISTRY: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase
  * HIV antibody, hepatitis GB surface antigen, hepatitis C antibody screens
  * URINALYSIS: by dipstick; full microscopic examination if dipstick positive
  * URINE DRUG SCREEN: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine

Exclusion Criteria

* Subjects with a recent history of drug or alcohol addiction or abuse.
* Subjects with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Subjects whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Subjects demonstrating a reactive screen for hepatitis B surface antigen, hepatitis C antibody or HIV antibody.
* Subjects demonstrating a positive drug abuse screen when screened for this study.
* Subjects with a history of allergic response(s) to pravastatin or related drugs.
* Subjects with a history of clinically significant allergies including drug allergies.
* Subjects with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Subjects who currently or report using tobacco products within 90 days of Period I dose administration.
* Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
* Subjects who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Subjects who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Subjects who report receiving any investigational drug within 28 days prior to Period I dosing.
* Subjects who report taking any systemic prescription medication in the 14 days prior to Period I dosing.
* Subjects who report an intolerance of direct venipuncture.
* Subjects who report consuming an abnormal diet during the 28 days prior to Period I dosing.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm D, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pravastatin (Test) First: Pravastatin 80 mg Tablet (test) dosed in first period followed by Pravachol® 80 mg Tablet (reference) dosed in second period
- Pravachol® (Reference) First: Pravachol® 80 mg Tablet (reference) dosed in first period followed by Pravastatin 80 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Pravastatin (Test) First | Pravachol® (Reference) First
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout: 7 Days
Arm/Group | Pravastatin (Test) First | Pravachol® (Reference) First
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Second Intervention
Arm/Group | Pravastatin (Test) First | Pravachol® (Reference) First
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pravastatin (Test) First | Pravachol® (Reference) First | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 8 | 6 | 14
  Hispanic | 0 | 1 | 1
  Black | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration - Pravastatin in Plasma
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 16 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Pravastatin: Pravastatin 80 mg Tablet (test) dosed in either period
- Pravachol®: Pravachol® 80 mg Tablet (reference) dosed in either period
Arm/Group | Pravastatin | Pravachol®
Number analyzed (Participants) | 15 | 15
ng/mL | 126.69 (60.95) | 130.64 (58.86)
Statistical Analysis 1: Comparison: Pravastatin vs Pravachol®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 98.45, 90% CI [80.08 to 121.03] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 16 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis. Data from one subject could not be included in the AUC0-inf calculation for Pravachol®.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Pravastatin | Pravachol®
Number analyzed (Participants) | 15 | 14
ng*h/mL | 273.32 (116.86) | 299.56 (121.83)
Statistical Analysis 1: Comparison: Pravastatin vs Pravachol®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 90.98, 90% CI [85.23 to 97.12] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 16 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Pravastatin | Pravachol®
Number analyzed (Participants) | 15 | 15
ng*h/mL | 241.29 (104.11) | 251.86 (111.26)
Statistical Analysis 1: Comparison: Pravastatin vs Pravachol®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Geometric Test/Ref Ratio x 100 = 96.30, 90% CI [85.34 to 108.66] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.